CLINICAL TRIAL: NCT06782958
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Characteristics of FHND1002 Granules After Single and Multiple Doses in Healthy Adult Volunteers
Brief Title: Safety, Tolerability, and Pharmacokinetics of FHND1002 Granules in Healthy Adults
Acronym: FHND1002-Ⅰ
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Chia Tai Fenghai Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FHND1002-I-01
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: FHND1002; Amyotrophic Lateral Sclerosis(ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Single dose (Experimental): Participants will receive a one-time dose (50 mg, 100 mg, 150 mg, 200 mg, or 250 mg) under fasting conditions or with a high-fat meal (for the 200 mg group).
  Interventions: Drug: 50mg FHND1002; Drug: 100mg FHND1002; Drug: 150 mg FHND1002; Drug: 200 mg FHND1002（fasting）; Drug: 250mg FHND1002; Drug: 200mg FHND1002(postprandial)
- Multiple dose (Experimental): Participants will receive daily doses (100 mg, 150 mg, or 200 mg) for 7 consecutive days under fasting conditions.
  Interventions: Drug: 100mg FHND1002; Drug: 150 mg FHND1002; Drug: 200 mg FHND1002（fasting）
- Placebo (Placebo Comparator): In the SAD phase, five dose groups (50 mg, 100 mg, 150 mg, 200 mg, and 250 mg) will be included, with 8 participants in each group (6 receiving FHND1002 and 2 receiving a placebo). Additionally, a food effect cohort (100 mg) will include 16 participants (14 receiving FHND1002 and 2 receiving a placebo), split into two groups to evaluate the impact of food under fasting and postprandial conditions.
  In the MAD phase, three dose groups (100 mg, 150 mg, and 200 mg) will be included, with 8 participants per group (6 receiving FHND1002 and 2 receiving a placebo). Participants will receive FHND1002 or placebo once daily under fasting conditions for 7 consecutive days.
  Interventions: Drug: 50mg FHND1002; Drug: 100mg FHND1002; Drug: 150 mg FHND1002; Drug: 200 mg FHND1002（fasting）; Drug: 250mg FHND1002; Drug: 200mg FHND1002(postprandial)

INTERVENTIONS:
Drug: 50mg FHND1002 — Participants will receive a daily oral dose of FHND1002 granules (50 mg) ,administered in the morning after fasting for at least 10 hours. The dose will be taken with 240 mL of water.
  Arms: Placebo; Single dose
Drug: 100mg FHND1002 — Participants will receive a daily oral dose of FHND1002 granules (100 mg) , administered in the morning after fasting for at least 10 hours. The dose will be taken with 240 mL of water.
Drug: 150 mg FHND1002 — Participants will receive a daily oral dose of FHND1002 granules (150 mg), administered in the morning after fasting for at least 10 hours. The dose will be taken with 240 mL of water.
Drug: 200 mg FHND1002（fasting） — Participants will receive a daily oral dose of FHND1002 granules (200 mg), administered in the morning after fasting for at least 10 hours. The dose will be taken with 240 mL of water.
Drug: 250mg FHND1002 — Participants will receive a daily oral dose of FHND1002 granules (250 mg), administered in the morning after fasting for at least 10 hours. The dose will be taken with 240 mL of water.
  Arms: Placebo; Single dose
Drug: 200mg FHND1002(postprandial) — Participants will receive a one-time dose (200 mg) under postprandial conditions
  Arms: Placebo; Single dose

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability, and pharmacokinetic (PK) profile of FHND1002 granules in healthy adult volunteers. The study will also assess how a high-fat meal affects the PK characteristics of FHND1002.

The main questions this study aims to answer are:

What are the safety and tolerability of FHND1002 granules when administered as single or multiple doses? What are the PK parameters of FHND1002, and what metabolites can be identified in humans?

Participants will:

Take FHND1002 granules or a placebo once daily, either as a single dose or for 7 consecutive days.

Attend regular clinic visits for checkups, tests, and blood sample collection. Undergo assessments, including monitoring for adverse events, physical exams, vital signs, ECGs, and laboratory tests.

DETAILED DESCRIPTION:
This study aims to evaluate the safety, tolerability, and pharmacokinetic (PK) profile of FHND1002 granules in healthy adult volunteers. The study is divided into two parts: a single ascending dose (SAD) phase and a multiple ascending dose (MAD) phase, with an additional evaluation of the effect of a high-fat meal on the PK characteristics of FHND1002.

The primary objectives of this study are:

To assess the safety and tolerability of FHND1002 granules following single and multiple doses in healthy volunteers.

To evaluate the impact of a high-fat meal on the PK profile of FHND1002 granules after a single oral dose.

The secondary objectives include:

To characterize the pharmacokinetic parameters of FHND1002 granules in healthy volunteers.

To identify and conduct preliminary research on drug metabolites in humans. This single-center, randomized, double-blind, placebo-controlled, single and multiple ascending dose Phase I clinical trial involves healthy adult volunteers. Based on preclinical pharmacodynamic, pharmacokinetic, and toxicological studies, as well as the formulation specifications of FHND1002 (25 mg and 100 mg), the maximum recommended starting dose for humans is set at 50 mg.

In the SAD phase, five dose groups (50 mg, 100 mg, 150 mg, 200 mg, and 250 mg) will be included, with 8 participants in each group (6 receiving FHND1002 and 2 receiving a placebo). Additionally, a food effect cohort (100 mg) will include 16 participants (14 receiving FHND1002 and 2 receiving a placebo), split into two groups to evaluate the impact of food under fasting and postprandial conditions.

In the MAD phase, three dose groups (100 mg, 150 mg, and 200 mg) will be included, with 8 participants per group (6 receiving FHND1002 and 2 receiving a placebo). Participants will receive FHND1002 or placebo once daily under fasting conditions for 7 consecutive days.

Throughout the study, participants will undergo regular assessments, including blood sample collection for PK analysis, adverse event (AE) monitoring, and evaluations such as physical exams, vital signs, ECGs, and laboratory tests. This study is expected to provide important data on the safety, tolerability, and pharmacokinetics of FHND1002, contributing to its further clinical development.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 and ≤45 years, regardless of gender.
* Male volunteers weigh ≥50 kg, and female volunteers weigh ≥45 kg, with a body mass index (BMI) between 19.0 and 26.0 kg/m² (inclusive).
* Medical history, physical examination, laboratory tests, and other assessments are normal or clinically insignificant, as determined by the investigator.
* Volunteers have no plans for pregnancy and voluntarily agree to use effective non-drug contraceptive measures (e.g., complete abstinence, condoms, sterilization) throughout the study and for three months after the last dose, with no plans for sperm or egg donation.
* Volunteers agree to comply with all study procedures and follow-up schedules and provide written informed consent.

Exclusion Criteria:

* History or presence of gastrointestinal, renal, hepatic, pulmonary, neurological, hematological, endocrine, oncological, immunological, psychiatric, or cardiovascular diseases that, in the investigator's opinion, may affect the safety of the volunteer or study results.
* History of severe allergies (e.g., angioedema or anaphylactic shock), hypersensitivity (e.g., to pollen or two or more drugs/foods), or known allergy to any components or excipients of the investigational drug.
* Use of any drugs that inhibit or induce hepatic drug metabolism (e.g., barbiturates, carbamazepine, phenytoin, corticosteroids) within 28 days before screening.
* Difficulty swallowing or a history of gastrointestinal diseases affecting drug absorption, digestive system surgeries (except for appendectomy, hemorrhoidectomy, or inguinal hernia repair), or known factors affecting pharmacokinetics.
* Underwent surgery within six months prior to screening or had surgery affecting drug absorption, distribution, metabolism, or excretion, as determined to be clinically significant by the investigator; or plans to undergo surgery during the study period.
* History of drug abuse, drug dependence, or a positive drug abuse screening result.
* Use of any prescription drugs, over-the-counter drugs, herbal medicines, or vitamins within 14 days prior to screening or within five half-lives of the drug before the first dose of the study drug (unless deemed irrelevant by the investigator).
* Participation in another clinical trial with drug administration within three months prior to the first dose of the study drug.
* Abnormal results in vital signs, electrocardiograms, ultrasounds, chest X-rays, or laboratory tests (e.g., blood routine, urinalysis, coagulation, blood biochemistry) deemed clinically significant by the investigator.
* Blood donation or other causes of blood loss exceeding 400 mL within three months prior to screening (excluding physiological blood loss in females).
* Difficulty with venous blood collection or a history of needle or blood phobia.
* Frequent alcohol consumption within three months prior to screening (defined as more than 14 units of alcohol per week, where 1 unit = 360 mL of beer, 45 mL of spirits with 40% alcohol, or 150 mL of wine), a positive alcohol breath test result, or inability to abstain from alcohol during the study.
* Vaccination within one month prior to the first dose or planned vaccination during the study or within one month after the study.
* Smoking more than five cigarettes per day within three months prior to screening or inability to abstain from tobacco use during the study.
* Excessive consumption of tea, coffee, or caffeine-containing beverages (more than 8 cups per day, where 1 cup = 250 mL) within three months prior to screening, consumption of specific foods (e.g., dragon fruit, mango, grapefruit) within 14 days prior to screening, or unwillingness to avoid caffeine-containing foods and beverages (e.g., tea, coffee, chocolate, cocoa), grapefruit products, or strenuous activities that may affect drug absorption, metabolism, or excretion during the study.
* Positive serological results for HBsAg, anti-HCV, anti-HIV, or TP-Ab at screening.
* Pregnant or breastfeeding female volunteers, or positive serum pregnancy test results.
* Male volunteers (or their partners) or female volunteers with plans for conception during the study period or within three months after study completion, or unwillingness to use non-drug contraceptive measures (e.g., complete abstinence, condoms, sterilization) during the study.
* Volunteers with specific dietary requirements (e.g., lactose intolerance) or unwillingness to adhere to the standardized diet provided during the study.
* Any other condition or factor that, in the investigator's judgment, renders the volunteer unsuitable for participation in the clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2025-03-03 (Estimated); Study Completion 2025-06-05 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 4 weeks
  This outcome measures the maximum observed plasma concentration of FHND1002 and its metabolites after single and multiple doses.
Time to Peak Plasma Concentration (Tmax) | 4 weeks
  This outcome evaluates the time required to reach maximum plasma concentration of FHND1002 and its metabolites.
Area Under the Curve from 0 to the Last Quantifiable Time Point (AUClast) | 4 weeks
  AUClast means Area Under the Concentration-Time Curve from 0 to the Last Quantifiable Time Point . This outcome assesses the total drug exposure up to the last measurable plasma concentration after single and multiple doses of FHND1002.
Area Under the Curve Over the Dosing Interval (AUCτ) | 4 weeks
  This outcome evaluates drug exposure during the dosing interval at steady state. τ means the dosing intervals.
Trough Concentration (Cmin) | 4 weeks
  The parameter is for multiple dose study. This outcome measures the minimum plasma concentration of FHND1002 and its metabolites before the next dose.
Average Plasma Concentration (Cavg) | 4 weeks
  The parameter is for multiple dose study. This outcome evaluates the average plasma concentration of FHND1002 during the dosing interval at steady state.
Accumulation Ratio (Rac) | 4 weeks
  Accumulation Ratio (Rac) is for Cmax and AUCτ. The outcome evaluates the accumulation of FHND1002 after multiple doses, calculated as the ratio of steady-state to single-dose parameters (e.g., Rac_Cmax, Rac_AUCτ).
Elimination Half-life (t1/2) | 4 weeks
  Elimination Half-life (t1/2) of FHND1002 assesses the time required for the plasma concentration of FHND1002 to decrease by half during the elimination phase.
Area Under the Curve from 0 to Infinity (AUC0-inf) | 4 weeks
  This outcome evaluates the total drug exposure from the time of dosing extrapolated to infinity for FHND1002 and its metabolites.
Incidence of Adverse Events(AEs) | 7 weeks
  This endpoint evaluates the safety of FHND1002 by monitoring the incidence of adverse events (AEs)
Incidence of Adverse Drug Reactions (ADRs) | 7 weeks
  This endpoint evaluates the safety of FHND1002 by monitoring the incidence of adverse drug reactions (ADRs),

SECONDARY OUTCOMES:
Coefficient of Variation (DF) of Pharmacokinetic Parameter | 4 weeks
  This outcome assesses the variability in pharmacokinetic parameters such as Cmax and AUCτ to understand inter- and intra-subject variability.
Apparent Clearance (CL/F) | 4 weeks
  This outcome evaluates the rate of drug clearance from the plasma after oral administration of FHND1002.
Apparent Volume of Distribution (Vz/F) | 4 weeks
  This outcome assesses the apparent volume of distribution of FHND1002 following oral administration, providing an estimate of drug distribution in the body.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Wang, Principal Investigator — LanZhou University
Locations (1):
- The first hospital of Lanzhou University, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No
Due to privacy and confidentiality concerns, individual participant data (IPD) will not be shared. The data contains sensitive health information that is protected by regulations, and sharing it may compromise participant confidentiality.

REFERENCES:
- [Background] Yu CH, Davidson S, Harapas CR, Hilton JB, Mlodzianoski MJ, Laohamonthonkul P, Louis C, Low RRJ, Moecking J, De Nardo D, Balka KR, Calleja DJ, Moghaddas F, Ni E, McLean CA, Samson AL, Tyebji S, Tonkin CJ, Bye CR, Turner BJ, Pepin G, Gantier MP, Rogers KL, McArthur K, Crouch PJ, Masters SL. TDP-43 Triggers Mitochondrial DNA Release via mPTP to Activate cGAS/STING in ALS. Cell. 2020 Oct 29;183(3):636-649.e18. doi: 10.1016/j.cell.2020.09.020. Epub 2020 Oct 7. PMID 33031745
- [Background] Watanabe H, Atsuta N, Hirakawa A, Nakamura R, Nakatochi M, Ishigaki S, Iida A, Ikegawa S, Kubo M, Yokoi D, Watanabe H, Ito M, Katsuno M, Izumi Y, Morita M, Kanai K, Taniguchi A, Aiba I, Abe K, Mizoguchi K, Oda M, Kano O, Okamoto K, Kuwabara S, Hasegawa K, Imai T, Kawata A, Aoki M, Tsuji S, Nakashima K, Kaji R, Sobue G. A rapid functional decline type of amyotrophic lateral sclerosis is linked to low expression of TTN. J Neurol Neurosurg Psychiatry. 2016 Aug;87(8):851-8. doi: 10.1136/jnnp-2015-311541. Epub 2016 Jan 8. PMID 26746183
- [Background] Xu L, Liu T, Liu L, Yao X, Chen L, Fan D, Zhan S, Wang S. Global variation in prevalence and incidence of amyotrophic lateral sclerosis: a systematic review and meta-analysis. J Neurol. 2020 Apr;267(4):944-953. doi: 10.1007/s00415-019-09652-y. Epub 2019 Dec 3. PMID 31797084
- [Background] Zhang J, Northoff G. Author Correction: Beyond noise to function: reframing the global brain activity and its dynamic topography. Commun Biol. 2022 Dec 21;5(1):1397. doi: 10.1038/s42003-022-04379-5. No abstract available. PMID 36543877
- [Background] Baughn MW, Melamed Z, Lopez-Erauskin J, Beccari MS, Ling K, Zuberi A, Presa M, Gonzalo-Gil E, Maimon R, Vazquez-Sanchez S, Chaturvedi S, Bravo-Hernandez M, Taupin V, Moore S, Artates JW, Acks E, Ndayambaje IS, Agra de Almeida Quadros AR, Jafar-Nejad P, Rigo F, Bennett CF, Lutz C, Lagier-Tourenne C, Cleveland DW. Mechanism of STMN2 cryptic splice-polyadenylation and its correction for TDP-43 proteinopathies. Science. 2023 Mar 17;379(6637):1140-1149. doi: 10.1126/science.abq5622. Epub 2023 Mar 16. PMID 36927019
- [Background] Fang MY, Markmiller S, Vu AQ, Javaherian A, Dowdle WE, Jolivet P, Bushway PJ, Castello NA, Baral A, Chan MY, Linsley JW, Linsley D, Mercola M, Finkbeiner S, Lecuyer E, Lewcock JW, Yeo GW. Small-Molecule Modulation of TDP-43 Recruitment to Stress Granules Prevents Persistent TDP-43 Accumulation in ALS/FTD. Neuron. 2019 Sep 4;103(5):802-819.e11. doi: 10.1016/j.neuron.2019.05.048. Epub 2019 Jul 1. PMID 31272829
- [Background] Piol D, Robberechts T, Da Cruz S. Lost in local translation: TDP-43 and FUS in axonal/neuromuscular junction maintenance and dysregulation in amyotrophic lateral sclerosis. Neuron. 2023 May 3;111(9):1355-1380. doi: 10.1016/j.neuron.2023.02.028. Epub 2023 Mar 23. PMID 36963381
- [Background] Mead RJ, Shan N, Reiser HJ, Marshall F, Shaw PJ. Amyotrophic lateral sclerosis: a neurodegenerative disorder poised for successful therapeutic translation. Nat Rev Drug Discov. 2023 Mar;22(3):185-212. doi: 10.1038/s41573-022-00612-2. Epub 2022 Dec 21. PMID 36543887
- [Background] Sheridan C. Unprecedented blood biomarker enables ALS drug approval. Nat Biotechnol. 2023 Jul;41(7):886-888. doi: 10.1038/s41587-023-01862-0. No abstract available. PMID 37386297
- [Background] Mullard A. ALS antisense drug falters in phase III. Nat Rev Drug Discov. 2021 Dec;20(12):883-885. doi: 10.1038/d41573-021-00181-w. No abstract available. PMID 34716445
- [Background] Todd TW, Petrucelli L. Modelling amyotrophic lateral sclerosis in rodents. Nat Rev Neurosci. 2022 Apr;23(4):231-251. doi: 10.1038/s41583-022-00564-x. Epub 2022 Mar 8. PMID 35260846